CLINICAL TRIAL: NCT05201599
Title: Treatment of Upper Urinary Tract Stones With a Diameter≤2cm by Flexible Ureteroscope With Intelligent Control of Renal Pelvic Pressure(FURL-ICP): a Multicenter, Parallel, Randomized Controlled Trial
Brief Title: Treatment of Upper Urinary Tract Stones With a Diameter≤2cm by Intelligent Pressure-controlled Flexible Ureteroscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other); Southern Medical University, China (Other); The Affiliated Ganzhou Hospital of Nanchang University (Other); The First Affiliated Hospital of Nanchang University (Other); Jiangxi Provincial People's Hopital (Other); The First Affiliated Hospital of Xiamen University (Other); Fujian Provincial Hospital (Other); First People's Hospital of Yulin (Other); Henan Provincial People's Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(49)2021
Record Dates: First submitted 2021-10-06; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Urinary Calculi
Keywords: upper urinary stone; flexible ureteroscope; vacuum suction; stone free rate
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: Patients with upper urinary stones ≤ 2cm in diameter will be assigned to intervention group (FURL-ICP group) or control group (f-URL) by a simple random sampling technique with a rate of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible ureteroscope with intelligent control of renal pelvic pressure(FURL-ICP) (Experimental): Patients will be placed in supine lithotomy position with 60-90° oblique on the affected side upward. A pressure measuring ureteral access sheath (UAS) (11-14Fr) is inserted into the proximal ureter along the guidewire without fluoroscopic guidance. The pressure sensory and suctioning channels are connected to the irrigation and suctioning platform.
  Interventions: Device: Flexible ureteroscope with intelligent control of renal pelvic pressure
- Traditional flexible ureteroscope(f-URL) (No Intervention): Each procedure is completed under general anesthesia in lithotomy position. A semi-rigid ureteroscopy is used to place a 0.032-inch guidewire. A pressure measuring ureteral access sheath (UAS) (11-14Fr) is inserted into the proximal ureter along the guidewire without fluoroscopic guidance. The irrigation and suctioning platform will be not used. A 7.5 Fr flexible ureteroscopy is used to break the stone with a holmium laser (fiber diameter 200 µm). A basket is used to remove the stone fragments. A 4-6Fr ureteral stent is left for 2 weeks after the operation. Stone composition is analyzed. If the UAS is failed to be placed, ureteral stent will be placed for 2 weeks and a second stage traditional f-URL will be performed.

INTERVENTIONS:
Device: Flexible ureteroscope with intelligent control of renal pelvic pressure — After adjusting the UAS in suitable position, the pressure sensory and suctioning channels are connected to the irrigation and suctioning platform. After being injected with water, a zero calibration is performed for the pressure sensory system. A fully automatic mode is selected on the platform. The perfusion flow is set between 50 to 150 mL/min. The RPP control value is set between -15 to -5 mmHg. The renal pelvic pressure alarm value is set between 20 to 30mmHg. During the operation, a holmium laser is used to break stones into powder (fiber diameter 200 µm), and the flexible ureteroscopy is moved back and forward slightly to suck out the stone particles inside the sheath gap. Particles larger than the sheath gap but smaller than the UAS is sucked out by intermittently withdrawing the flexible ureteroscope without basket.
  Arms: Flexible ureteroscope with intelligent control of renal pelvic pressure(FURL-ICP)

SUMMARY:
The aim of this trial is to compare the efficacy and safety of flexible ureteroscope with intelligent control of renal pelvic pressure (FURL-ICP) and traditional flexible ureteroscope(f-URL) in the treatment of upper urinary stones ≤ 2cm in diameter. It is designed as a multicenter, parallel randomized controlled trial with two arms. At least 449 patients with upper urinary stones ≤ 2cm in diameter will be invited to participant in this study. Patients will be assigned to intervention group (FURL-ICP group) or control group (f-URL) by a simple random sampling technique with a rate of 1:1. The baseline of participants include demographic data, urine analysis, blood cell analysis, blood biochemical analysis, and urinary computer tomography (CT) with a slice thickness of 2mm. The primary outcomes are postoperative stone-free rate (SFR) of one month by CT scan and postoperative fever rate (body temperature > 38.5 ℃ within 3 days after operation). Secondary outcomes include operating time, degree of ureteral injury, SFR of one day.

DETAILED DESCRIPTION:
1. Background Urinary stone is a common disease with a prevalence rate of 5-15%. It has a recurrence rate of 50% for 5-10 years, and about 75% for 20 years. It is a heavy healthy burden to the population. Flexible ureteroscope lithotripsy(f-URL) is a first-line treatment for renal stone ≤ 2cm in diameter. It has the advantage of less trauma, low complications and fast recovery. It is also suitable for upper ureteral calculi, residual calculi after percutaneous nephrolithotomy (PCNL) It can also be combined with PCNL for the treatment of complex renal calculi.

   The postoperative stone free rate of f-URL varies drastically due to different sizes of residual stone. The Chinese consensus of flexible ureteroscopy recommended that stone ≤ 4mm in diameter should be considered as clinical insignificant residual stone. When residual stone was defined as ≤ 3mm, the stone free rate for one-month was 90% of renal stones ≤ 20 mm, and was 74.4% for stone of 10-25 mm. It would not cause significant symptoms when the residual stone ≤ 2 mm. Based on this definition, Fatih A's randomized trial showed that the stone free rate of f-URL for renal calculi ≤ 20 mm was 85.7%. It was only 30% for stone > 20 mm of single procedure，86.6% of secondary procedure, and 100% for tertiary procedure. When the residual stone was defined as ≤ 1 mm, the stone free rate of f-URL was 64.7% for a single procedure, 92% for secondary procedure, and the overall stone free rate was 85.1% and 100% for stone > 20 mm and ≤ 20 mm respectively by a retrospective study. When the stone free rate was defined as complete stone clearance, it was 71% after one month of single f-URL for renal stone >30mm .

   Postoperative infection is a common complication of f-URL. The key point to avoid postoperative infection includes to treat urinary infection, to keep a low flow perfusion and renal pelvic pressure (RPP) during operation, and to control the operation time. The renal pelvic pressure depends on the size of ureteral sheath and flexible ureteroscope, the flow of perfusion and outflow of traditional f-URL. It is difficult to realize real-time monitoring and regulation of renal pelvic pressure during the operation.

   To realize a high stone free rate and a low postoperative infection rate of f-URL, a new system named flexible ureteroscope with intelligent control of renal pelvic pressure (FURL-ICP) is designed and used. It has an irrigation and suctioning control platform, uses a ureteral access sheath with a pressure-sensitive tip, enables regulation of the infusion flow precisely, and controls the vacuum suctioning by computerized real-time recording and monitoring of RPP. A stable RPP is kept within a pre-set safe range by pressure feedback technology. The stone power could be sucked out during operation. Previous data showed that postoperative stone free rate was 90% for one day, and 95.6% for one month after operation respectively, and the overall complication rate was 14.4%. The aim of this study is to compare the efficacy and safety for FURL-ICP and f-URL in the treatment of upper urinary calculi with diameter ≤ 2cm.
2. Objective To compare the efficacy and safety of FURL-ICP and traditional FURL for the treatment of ≤ 2cm upper urinary stones.
3. Trial Design and Participants The trial is designed as a multicenter, parallel, randomized controlled trial with two arms. Patients will be recruited from 12 Chinese tertiary medical centers. Each participating center performed >50 f-URLs per month. Patients with upper urinary tract stones scheduled for f-URL will be invited in this study.
4. Randomization and masking Central randomized allocation will be used without stratification. Participants will be assigned by a simple random sampling technique with a rate of 1:1. A randomization list is generated by a statistician and securely stored at a password-protected computer of the sponsor's center. Only one protocol-blinded coordinator will know the password and reveal the assignments in sequence to each center. The allocation is revealed before the surgery day. One-side superiority test is designed to compare the efficacy and safety of FURL-ICP and f-URL.
5. Sample size Sample size is estimated by SFR of one month for f-URL. Complete stone free is defined as residual stone ≤ 2mm in diameter. The SFRs of FURL-ICP and traditional f-URL are presumed to be 90% (PT) and 75% (PC) respectively, based on previous data. 5% is considered as an inferior margin. The sample size is calculated with the formulas of a one-side superiority test comparing two proportions. The minimum sample size for each group was 224, and at least 449 cases are needed in the study. (https://www.cnstat.org/statx/compute.html).
6. Intervention methods:

（1）Operation methods of intervention group(FURL-ICP)： Each procedure is completed under general anesthesia in supine lithotomy position with 60-90° oblique on the affected side upward. A semi-rigid ureteroscopy is used to check the urinary tract system and to place a 0.032-inch guidewire. A pressure measuring ureteral access sheath (UAS) (11/13.8Fr) is inserted into the proximal ureter along the guidewire without fluoroscopic guidance. A 7.5 Fr flexible ureteroscopy is used to check the delivery location of the UAS, mucosa of renal pelvis and ureter. After adjusting the UAS in suitable position, the pressure sensory and suctioning channels are connected to the irrigation and suctioning platform. After being injected with water, a zero calibration is performed for the pressure sensory system. A fully automatic mode is selected on the platform. The perfusion flow is set between 50 to 150 mL/min. The RPP control value is set between -15 to -5 mmHg. The renal pelvic pressure alarm value is set between 20 to 30mmHg. During the operation, a holmium laser is used to break stones into powder (fiber diameter 200 µm), and the flexible ureteroscopy is moved back and forward slightly to suck out the stone particles inside the sheath gap. Particles larger than the sheath gap but smaller than the UAS is sucked out by intermittently withdrawing the flexible ureteroscopy without basketing. A 4-6Fr ureteral stent is left for 2 weeks after the operation. Stone composition is analyzed. If the UAS is failed to be placed, ureteral stent will be placed for 2 weeks and a second stage FURL-ICP will be performed.

（2）Operation methods of control group（traditional f-URL）： Each procedure is completed under general anesthesia in lithotomy position. A semi-rigid ureteroscopy is used to place a 0.032-inch guidewire. A pressure measuring ureteral access sheath (UAS) (11/13.8Fr) is inserted into the proximal ureter along the guidewire without fluoroscopic guidance. The irrigation and suctioning platform will be not used. A 7.5 Fr flexible ureteroscopy is used to break the stone with a holmium laser (fiber diameter 200 µm). A basket is used to remove the stone fragments. A 4-6Fr ureteral stent is left for 2 weeks after the operation. Stone composition is analyzed. If the UAS is failed to be placed, ureteral stent will be placed for 2 weeks and a second stage traditional f-URL will be performed.

ELIGIBILITY:
Inclusion Criteria:

* The diameter of single stone or cumulative maximum diameter for multiple stones is less than or equal to 2cm
* American Society of Anesthesiology scores of 1to 2
* All patients participate in this study voluntarily and signed informed consent

Exclusion Criteria:

* Uncontrolled urinary tract infection
* Patients with pyonephrosis are found during operation
* The patients with abnormal anatomy (heterotopic kidney, horseshoe kidney, duplicate kidney), ureteral stricture, urethral stricture and urinary diversion
* Severe hydronephrosis
* Renal function was decompensated (serum creatinine > 178 μmol/L)
* Severe systemic hemorrhagic disease
* Patients who underwent bilateral surgery at the same time
* Severe deformity of hip joint and difficult position

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Stone free rate for one month | One month after surgery
  Stone free rate for one month after surgery by CT scan with a thickness of 2mm.

SECONDARY OUTCOMES:
Stone free rate for one day | One day after surgery
  Stone free rate for one day after surgery by X-ray.
Postoperative fever rate | Within 3 days after operation
  Postoperative fever rate (body temperature > 38.5°C within 3 days after operation
Operating time | During the operation
  Operating time
Degree of ureteral injury | During the operation
  Degree of ureteral injury

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, Doctor, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Affiliated Ganzhou Hospital of Nanchang University (Ganzhou People's Hospital), Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
When the study is finished, we will shared data with other researchers.

REFERENCES:
- [Result] Zeng G, Mai Z, Xia S, Wang Z, Zhang K, Wang L, Long Y, Ma J, Li Y, Wan SP, Wu W, Liu Y, Cui Z, Zhao Z, Qin J, Zeng T, Liu Y, Duan X, Mai X, Yang Z, Kong Z, Zhang T, Cai C, Shao Y, Yue Z, Li S, Ding J, Tang S, Ye Z. Prevalence of kidney stones in China: an ultrasonography based cross-sectional study. BJU Int. 2017 Jul;120(1):109-116. doi: 10.1111/bju.13828. Epub 2017 Mar 21. PMID 28236332
- [Result] Moe OW. Kidney stones: pathophysiology and medical management. Lancet. 2006 Jan 28;367(9507):333-44. doi: 10.1016/S0140-6736(06)68071-9. PMID 16443041
- [Result] Farhan M, Nazim SM, Salam B, Ather MH. Prospective evaluation of outcome of percutaneous nephrolithotomy using the 'STONE' nephrolithometry score: A single-centre experience. Arab J Urol. 2015 Dec;13(4):264-9. doi: 10.1016/j.aju.2015.07.006. Epub 2015 Aug 29. PMID 26609445
- [Result] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Result] Khan SR, Pearle MS, Robertson WG, Gambaro G, Canales BK, Doizi S, Traxer O, Tiselius HG. Kidney stones. Nat Rev Dis Primers. 2016 Feb 25;2:16008. doi: 10.1038/nrdp.2016.8. PMID 27188687
- [Result] Trinchieri A, Ostini F, Nespoli R, Rovera F, Montanari E, Zanetti G. A prospective study of recurrence rate and risk factors for recurrence after a first renal stone. J Urol. 1999 Jul;162(1):27-30. doi: 10.1097/00005392-199907000-00007. PMID 10379732
- [Result] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Result] Guler Y, Erbin A, Ozmerdiven G, Yazici O. Comparison of Retrograde Intrarenal Surgery and Laparoscopic Surgery in the Treatment of Proximal Ureteral and Renal Pelvic Stones Greater than 15 mm. Folia Med (Plovdiv). 2020 Sep 30;62(3):490-496. doi: 10.3897/folmed.62.e48934. PMID 33009767
- [Result] Resorlu B, Unsal A, Ziypak T, Diri A, Atis G, Guven S, Sancaktutar AA, Tepeler A, Bozkurt OF, Oztuna D. Comparison of retrograde intrarenal surgery, shockwave lithotripsy, and percutaneous nephrolithotomy for treatment of medium-sized radiolucent renal stones. World J Urol. 2013 Dec;31(6):1581-6. doi: 10.1007/s00345-012-0991-1. Epub 2012 Nov 22. PMID 23179732
- [Result] Cvetkovic T, Kameric-Buljina M. [Comparative "in vitro" examination of permeability of rebasing made of phosphate cement and tubulitec aiming at chemical protection of dental pulp]. Stomatol Vjesn. 1986;15(1-2):23-7. No abstract available. Croatian. PMID 3484138
- [Result] Javanmard B, Kashi AH, Mazloomfard MM, Ansari Jafari A, Arefanian S. Retrograde Intrarenal Surgery Versus Shock Wave Lithotripsy for Renal Stones Smaller Than 2 cm: A Randomized Clinical Trial. Urol J. 2016 Oct 10;13(5):2823-2828. PMID 27734422
- [Result] Hussain M, Acher P, Penev B, Cynk M. Redefining the limits of flexible ureterorenoscopy. J Endourol. 2011 Jan;25(1):45-9. doi: 10.1089/end.2010.0236. Epub 2010 Nov 4. PMID 21050026
- [Result] Karakoyunlu N, Goktug G, Sener NC, Zengin K, Nalbant I, Ozturk U, Ozok U, Imamoglu A. A comparison of standard PCNL and staged retrograde FURS in pelvis stones over 2 cm in diameter: a prospective randomized study. Urolithiasis. 2015 Jun;43(3):283-7. doi: 10.1007/s00240-015-0768-2. Epub 2015 Apr 3. PMID 25838180
- [Result] Akbulut F, Kucuktopcu O, Kandemir E, Sonmezay E, Simsek A, Ozgor F, Binbay M, Muslumanoglu AY, Gurbuz G. Comparison of flexible ureterorenoscopy and mini-percutaneous nephrolithotomy in treatment of lower calyceal stones smaller than 2 cm. Ren Fail. 2016;38(1):163-7. doi: 10.3109/0886022X.2015.1128792. Epub 2016 Jan 4. PMID 26727075
- [Result] Yanaral F, Ozgor F, Kucuktopcu O, Sarilar O, Ayranci A, Savun M, Yuksel B, Binbay M. Comparison of Flexible Ureterorenoscopy and Mini Percutaneous Nephrolithotomy in the Management of Multiple Renal Calculi in 10-30 mm Size. Urol J. 2019 Aug 18;16(4):326-330. doi: 10.22037/uj.v0i0.3310. PMID 30334245
- [Result] Saad KS, Youssif ME, Al Islam Nafis Hamdy S, Fahmy A, El Din Hanno AG, El-Nahas AR. Percutaneous Nephrolithotomy vs Retrograde Intrarenal Surgery for Large Renal Stones in Pediatric Patients: A Randomized Controlled Trial. J Urol. 2015 Dec;194(6):1716-20. doi: 10.1016/j.juro.2015.06.101. Epub 2015 Jul 10. PMID 26165587
- [Result] Deng X, Song L, Xie D, Fan D, Zhu L, Yao L, Wang X, Liu S, Zhang Y, Liao X, Liu S, Peng Z, Hu M, Zhu X, Huang J, Liu T, Du C, Guo S, Yang Z, Peng G, Ye Z. A Novel Flexible Ureteroscopy with Intelligent Control of Renal Pelvic Pressure: An Initial Experience of 93 Cases. J Endourol. 2016 Oct;30(10):1067-1072. doi: 10.1089/end.2015.0770. Epub 2016 Sep 28. PMID 27558001
- [Result] Chen H, Qiu X, Du C, Xie D, Liu T, Wang G, Song L. The Comparison Study of Flexible Ureteroscopic Suctioning Lithotripsy With Intelligent Pressure Control Versus Minimally Invasive Percutaneous Suctioning Nephrolithotomy in Treating Renal Calculi of 2 to 3 cm in Size. Surg Innov. 2019 Oct;26(5):528-535. doi: 10.1177/1553350619849782. Epub 2019 May 26. PMID 31130072
- [Derived] Deng X, Chen Y, Zhai Q, Song L, Du C, Tan W. Fluid absorption during flexible ureteroscopy with intelligent control of renal pelvic pressure: a randomized controlled trial. World J Urol. 2024 May 17;42(1):331. doi: 10.1007/s00345-024-05036-8. PMID 38758400
- Available data/document: Study Protocol: zxt4 — https://pan.baidu.com/s/1PNKfPWrpeJtodX1RwH8k-w